CLINICAL TRIAL: NCT02408237
Title: Development of Apparatus of Transcranial Direct Current Stimulation (tDCS) for Domiciliary Use
Brief Title: Transcranial Direct Current Stimulation Apparatus for Domiciliary Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Wolnei Caumo, Wolnei Caumo, MD, PhD, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Device Feasibility
Other Study IDs: 14-0281
Record Dates: First submitted 2015-02-25; First posted 2015-04-03 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-03

CONDITIONS: Transcranial Direct Current Stimulation; Healthy Participants
Keywords: Transcranial direct current stimulation (tDCS); tDCS for domiciliary use; Healthy Participants
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS Ambulatory & Sham (Active Comparator): Active tDCS Ambulatory: 1 mA of current of active tDCS applied for 20 minutes, single session of stimulation. Sham tDCS Ambulatory: applied for 20 minutes, single session of stimulation.
  Interventions: Device: Active tDCS Ambulatory; Device: Sham tDCS Ambulatory
- tDCS home use & Sham (Active Comparator): Active tDCS home use: 11 active tDCS sessions: single session in the hospital and the remaining 10 in the subject's home, with duration of each active tDCS session of 20 min. Sham tDCS home use: 11 sessions of tDCS: single session in the hospital and the remaining 10 in the subject's home, with duration of each sham tDCS session of 20 min.
  Interventions: Device: Active tDCS Home use; Device: Sham tDCS Home use

INTERVENTIONS:
Device: Active tDCS Ambulatory — Procedure begins with the placement of an anode electrode placed on the primary motor cortex (cortex contralateral to the dominant) and the cathode is placed on the contralateral supraorbital region. It is used 1mA direct current transcranial stimulation applied for 20 minutes. Will be held a single session of stimulation. The total time, with initial assessment, tDCS session and final evaluation will be approximately 4 hours.
  Other Names: Transcranial Direct Current Stimulation
  Arms: tDCS Ambulatory & Sham
Device: Sham tDCS Ambulatory — In sham group, we follow the same procedure and time as the active tDCS ambulatory protocol, but the device will be in the mode sham (inactive). The current is only applied for 30 seconds, so subjects feel a sense of the initial stimulation, but not the remainder receive current. In this group one session will also be held. The total time, with initial assessment, tDCS session and final evaluation will be approximately 4 hours.
  Other Names: Transcranial Direct Current Stimulation
  Arms: tDCS Ambulatory & Sham
Device: Active tDCS Home use — The procedure and stimulation time is exactly the same that Active tDCS - ambulatory use, but will use the apparatus for domestic use. Will be explained to the participant as placement of the cap and the device management. This group will be made 11 sessions of tDCS, the first held in the Hospital, with supervision of the researcher. The remaining 10 will be held in the participant's home. The total time of the first meeting, with initial assessment, tDCS session and final evaluation will be around 4 hours. The time of last evaluation is approximately 1 hour.
  Other Names: Transcranial Direct Current Stimulation
  Arms: tDCS home use & Sham
Device: Sham tDCS Home use — The procedure and stimulation time is exactly the same that Active tDCS - ambulatory use, but will use the apparatus for domestic use. In sham group, we follow the same procedure and time as the active tDCS protocol, but the device will be in the sham mode (inactive). The total time of the first meeting, with initial assessment, tDCS session and final evaluation will be around 4 hours. The time of last evaluation is approximately 1 hour.
  Other Names: Transcranial Direct Current Stimulation
  Arms: tDCS home use & Sham

SUMMARY:
Neuromodulation is characterized as a technique whose principle neurostimulation to produce inhibition or cortical arousal. The tDCS (transcranial direct current stimulation) is a noninvasive brain stimulation method used to modulate cortical excitability using low intensity direct current (1-2mA) directed to the scalp via cathodes and anodes electrodes; the current reaches the cortex, producing hyperpolarization or depolarization of the axonal membrane potential. Evidence has shown that this method is presented as a technique that can alter cortical and subcortical neural networks. This technique has been used to treat psychiatric disorders such as depression, acute mania, bipolar affective disorder panic, hallucinations, obsessive compulsive disorder, schizophrenia, withdrawal, rehabilitation after-stroke and pain syndromes such as neuropathic pain, migraine, pancreatitis chronic pain and fibromyalgia. It is low-cost technique, with virtually no side effects and carries the therapeutic effect by neuromodulatory pathways by distinct pathways activated by the drugs. In this scenario falls within the importance of developing devices for home use, inexpensive, and easy to use so as to maintain the benefits observed in previous studies. The tDCS is presented as a non-pharmacological option that may be offered in this context in society. It is noteworthy that, if the benefit is demonstrated, the impact will be of great importance to patients and to society, since these are focal techniques and low cost. Because they have no focal adverse effects of conventional drug treatments. Additionally, can be constituted as technical additive to pharmacotherapy in so much pain as in the treatment of other neuropsychiatric disorders. Therefore, further studies should be encouraged to increase knowledge of their effects and mechanisms involved. If the effectiveness of this method for home use is confirmed, the therapeutic impact will undoubtedly be of great importance. However, to make this project come true, the investigators depend on support for the development and validation of tDCS device for home use, so allowing the qualified knowledge can be applied to the clinical setting, as well as advance the development of this area of neuroscience in Brazil. Therefore, the aim of this study is to develop tDCS device for home use.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged between 18 and 40 years.
* Higher education (college graduates in progress or completed).

Exclusion Criteria:

* Subject left-handed.
* History of neurological disease.
* History of endocrine disease.
* History of psychiatric disorder.
* History of sleep disorders (apnea, hypersomnia, insomnia, sleepwalking ...).
* Chronic pain.
* Chronic inflammatory and oncological diseases.
* Systemic arterial hypertension; ischemic heart disease.
* Kidney and liver failure.
* Regular use of steroids and non-steroids anti inflammatory, opioids and non-opioids, psychotropics, anticonvulsants, alpha and beta-blockers.
* Regular use of drugs, alcohol and tobacco.
* History of brain surgery, tumor, stroke or intracranial implantation of metal (or not implemented).
* Subjects who do not understand Portuguese.
* Body mass index greater than 29.9.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
Cortical excitability on the transcranial magnetic stimulation (TMS) | 2 days
  Evaluation of the variation in cortical excitability parameters pre and post application of tDCS: Motor evoked potential (MEP); Motor threshold (MT); intracortical facilitation, intracortical inhibition, silent period (SP).

SECONDARY OUTCOMES:
Serum levels of Brain Derived Neurotrophic Factor (BDNF) | 2 days
  Measurement of serum levels of BDNF pre and post application of tDCS.
Pressure pain threshold | 2 days
  Measurement of pressure pain threshold pre and post application of tDCS.
Heat pain threshold | 2 days
  Measurement of heat pain threshold pre and post application of tDCS, with quantitative sensory test (QST).
Conditional pain modulation (CPM) | 2 days
  Assessment of conditional pain modulation pre and post application of tDCS, with cold and hot threshold.
Number of participants with adverse events after use tDCS | 10 days
  Assessment of adverse events after use of Transcranial Direct Current Stimulation Apparatus for Domiciliary Use.

CONTACTS AND LOCATIONS:
Overall Officials: Wolnei Caumo, PhD, Study Director — +55513359808
Locations (1):
- Fabiana Carvalho, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stagg CJ, Nitsche MA. Physiological basis of transcranial direct current stimulation. Neuroscientist. 2011 Feb;17(1):37-53. doi: 10.1177/1073858410386614. PMID 21343407
- [Background] Nitsche MA, Paulus W. Sustained excitability elevations induced by transcranial DC motor cortex stimulation in humans. Neurology. 2001 Nov 27;57(10):1899-901. doi: 10.1212/wnl.57.10.1899. PMID 11723286
- [Background] Nitsche MA, Fricke K, Henschke U, Schlitterlau A, Liebetanz D, Lang N, Henning S, Tergau F, Paulus W. Pharmacological modulation of cortical excitability shifts induced by transcranial direct current stimulation in humans. J Physiol. 2003 Nov 15;553(Pt 1):293-301. doi: 10.1113/jphysiol.2003.049916. Epub 2003 Aug 29. PMID 12949224
- [Background] Martin DM, Alonzo A, Ho KA, Player M, Mitchell PB, Sachdev P, Loo CK. Continuation transcranial direct current stimulation for the prevention of relapse in major depression. J Affect Disord. 2013 Jan 25;144(3):274-8. doi: 10.1016/j.jad.2012.10.012. Epub 2012 Nov 10. PMID 23146197
- [Background] Valiengo L, Bensenor IM, Goulart AC, de Oliveira JF, Zanao TA, Boggio PS, Lotufo PA, Fregni F, Brunoni AR. The sertraline versus electrical current therapy for treating depression clinical study (select-TDCS): results of the crossover and follow-up phases. Depress Anxiety. 2013 Jul;30(7):646-53. doi: 10.1002/da.22079. Epub 2013 Apr 26. PMID 23625554
- [Background] DaSilva AF, Volz MS, Bikson M, Fregni F. Electrode positioning and montage in transcranial direct current stimulation. J Vis Exp. 2011 May 23;(51):2744. doi: 10.3791/2744. PMID 21654618
- [Background] Iyer MB, Mattu U, Grafman J, Lomarev M, Sato S, Wassermann EM. Safety and cognitive effect of frontal DC brain polarization in healthy individuals. Neurology. 2005 Mar 8;64(5):872-5. doi: 10.1212/01.WNL.0000152986.07469.E9. PMID 15753425
- [Background] Nitsche MA, Cohen LG, Wassermann EM, Priori A, Lang N, Antal A, Paulus W, Hummel F, Boggio PS, Fregni F, Pascual-Leone A. Transcranial direct current stimulation: State of the art 2008. Brain Stimul. 2008 Jul;1(3):206-23. doi: 10.1016/j.brs.2008.06.004. Epub 2008 Jul 1. PMID 20633386
- [Background] Priori A. Brain polarization in humans: a reappraisal of an old tool for prolonged non-invasive modulation of brain excitability. Clin Neurophysiol. 2003 Apr;114(4):589-95. doi: 10.1016/s1388-2457(02)00437-6. PMID 12686266
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Background] Lang N, Siebner HR, Ward NS, Lee L, Nitsche MA, Paulus W, Rothwell JC, Lemon RN, Frackowiak RS. How does transcranial DC stimulation of the primary motor cortex alter regional neuronal activity in the human brain? Eur J Neurosci. 2005 Jul;22(2):495-504. doi: 10.1111/j.1460-9568.2005.04233.x. PMID 16045502
- [Background] Medeiros LF, de Souza IC, Vidor LP, de Souza A, Deitos A, Volz MS, Fregni F, Caumo W, Torres IL. Neurobiological effects of transcranial direct current stimulation: a review. Front Psychiatry. 2012 Dec 28;3:110. doi: 10.3389/fpsyt.2012.00110. eCollection 2012. PMID 23293607
- [Background] Garcia-Larrea L, Peyron R, Mertens P, Gregoire MC, Lavenne F, Le Bars D, Convers P, Mauguiere F, Sindou M, Laurent B. Electrical stimulation of motor cortex for pain control: a combined PET-scan and electrophysiological study. Pain. 1999 Nov;83(2):259-73. doi: 10.1016/s0304-3959(99)00114-1. PMID 10534598
- [Background] Fregni F, Boggio PS, Lima MC, Ferreira MJ, Wagner T, Rigonatti SP, Castro AW, Souza DR, Riberto M, Freedman SD, Nitsche MA, Pascual-Leone A. A sham-controlled, phase II trial of transcranial direct current stimulation for the treatment of central pain in traumatic spinal cord injury. Pain. 2006 May;122(1-2):197-209. doi: 10.1016/j.pain.2006.02.023. Epub 2006 Mar 27. PMID 16564618
- [Background] Fregni F, Gimenes R, Valle AC, Ferreira MJ, Rocha RR, Natalle L, Bravo R, Rigonatti SP, Freedman SD, Nitsche MA, Pascual-Leone A, Boggio PS. A randomized, sham-controlled, proof of principle study of transcranial direct current stimulation for the treatment of pain in fibromyalgia. Arthritis Rheum. 2006 Dec;54(12):3988-98. doi: 10.1002/art.22195. PMID 17133529
- [Background] Silva G, Miksad R, Freedman SD, Pascual-Leone A, Jain S, Gomes DL, Amancio EJ, Boggio PS, Correa CF, Fregni F. Treatment of cancer pain with noninvasive brain stimulation. J Pain Symptom Manage. 2007 Oct;34(4):342-5. doi: 10.1016/j.jpainsymman.2007.06.002. No abstract available. PMID 17903664
- [Background] Fregni F, Freedman S, Pascual-Leone A. Recent advances in the treatment of chronic pain with non-invasive brain stimulation techniques. Lancet Neurol. 2007 Feb;6(2):188-91. doi: 10.1016/S1474-4422(07)70032-7. PMID 17239806
- [Background] Drewes AM, Gregersen H, Arendt-Nielsen L. Experimental pain in gastroenterology: a reappraisal of human studies. Scand J Gastroenterol. 2003 Nov;38(11):1115-30. doi: 10.1080/00365520310004399. No abstract available. PMID 14686714
- [Background] Boggio PS, Zaghi S, Lopes M, Fregni F. Modulatory effects of anodal transcranial direct current stimulation on perception and pain thresholds in healthy volunteers. Eur J Neurol. 2008 Oct;15(10):1124-30. doi: 10.1111/j.1468-1331.2008.02270.x. Epub 2008 Aug 20. PMID 18717717
- [Background] Liebetanz D, Koch R, Mayenfels S, Konig F, Paulus W, Nitsche MA. Safety limits of cathodal transcranial direct current stimulation in rats. Clin Neurophysiol. 2009 Jun;120(6):1161-7. doi: 10.1016/j.clinph.2009.01.022. Epub 2009 Apr 28. PMID 19403329
- [Background] Bikson M, Datta A, Elwassif M. Establishing safety limits for transcranial direct current stimulation. Clin Neurophysiol. 2009 Jun;120(6):1033-4. doi: 10.1016/j.clinph.2009.03.018. Epub 2009 Apr 24. No abstract available. PMID 19394269
- [Background] Minhas P, Bansal V, Patel J, Ho JS, Diaz J, Datta A, Bikson M. Electrodes for high-definition transcutaneous DC stimulation for applications in drug delivery and electrotherapy, including tDCS. J Neurosci Methods. 2010 Jul 15;190(2):188-97. doi: 10.1016/j.jneumeth.2010.05.007. Epub 2010 May 19. PMID 20488204
- [Background] Rolke R, Magerl W, Campbell KA, Schalber C, Caspari S, Birklein F, Treede RD. Quantitative sensory testing: a comprehensive protocol for clinical trials. Eur J Pain. 2006 Jan;10(1):77-88. doi: 10.1016/j.ejpain.2005.02.003. PMID 16291301